CLINICAL TRIAL: NCT05809479
Title: NICE - Nutritional Impact on Immunological Maturation During Childhood in Relation to the Environment
Acronym: NICE
Status: Active, not recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Göteborg University (Other); Chalmers University of Technology (Other); Karolinska Institutet (Other); Region Norrbotten (Unknown); The Swedish Research Council (Other Government); Forte (Industry); The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Dnr 2013-18-31M
Record Dates: First submitted 2023-03-14; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Chronic Diseases in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, faeces, blood, placenta, hair, breast milk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Role of the exposome on allergy, caries, and neurophysiological development in childhood.

DETAILED DESCRIPTION:
Role of the exposome and epigenetics on allergy, caries, and neurophysiological development in childhood as studied in a birth cohort of 650 trioses. The exposome includes repeated measures of nutrition, micronutritients, microbiota, toxic agents and the clinical outcomes, diagnoses of allergy, caries and neurophysiological functions/dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Born at Sunderby hospital, Region Norrbotten, during time period 2015-2018

Exclusion Criteria:

* Parents not able to speak or write Swedish

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 650 families (mother/father/child).
Sampling Method: Non-Probability Sample
Enrollment: 1950 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with excema | Outcome at one year
  Excema
Number of participants with food allergy | Outcome at one year
  Food allergy
Number of participants with frhino-conjuctivitis | Outcome at one year
  Rhino-conjunctivitis
Number of participants with asthma | Outcome at one year
  Asthma
Number of participants with excema | Outcome at four years
  Excema
Number of participants with food allergy | Outcome at four years
  Food allergy
Number of participants with rhino-conjunctivitis | Outcome at four years
  Rhino-conjuctivitis
Number of participants with asthma | Outcome at four years
  Asthma
Number of participants with excema | Outcome at six years
  Excema
Number of participants with food allergy | Outcome at six years
  Food allergy
Number of participants with rhino-conjunctivitis | Outcome at six years
  Rhino-conjunctivitis
Number of participants with asthma | Outcome at six years
  Asthma
Numbers of caries lesions (DeMFS = decayed, enamel included, missed, filled, tooth surfaces, in each child | Outcome at four years
  Cariesfree individuals have a DeMFS = 0 and increasing scores means increasing degree of caries. Maximum DeMFS = 148, minumum DeMFS = 0.
Child cognition as measured by Wechsler Preschool and Primary Scale of Intelligence | Outcome at four years
  Cognitive development will be tested face-to-face with Wechsler Preschool and Primary Scale of Intelligence. Increasing scores means increasing intelligence.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sandin, Ass Prof, Principal Investigator — Umeå University
Locations (1):
- Sunderby Hospital, Luleå, Norrbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No